CLINICAL TRIAL: NCT07077382
Title: Pneumoconiosis and Dust Exposure China Cohort
Acronym: PANDECT
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: KaiLuan General Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Weifang Respiratory Disease Hospital (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Hunan Prevention and Treatment Institute for Occupational Diseases, China (Unknown); The first affiliated hospital of chongqing medical and pharmaceutical college (Unknown); Centers for Disease Control and Prevention, China (Other Government); Shandong Gold Mining Company Occupational Disease Precention Hospital (Unknown); Shandong Province Hospital of occupational diseases (Unknown); The Second Hospital of Heilongjiang Province (Unknown)
Responsible Party: Principal Investigator, Dai Huaping, Chief physician, China-Japan Friendship Hospital
Other Study IDs: ChinaJapanFH005
Record Dates: First submitted 2025-06-23; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pneumoconiosis
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

GROUPS / COHORTS (3):
- Patients with pneumoconiosis: This group is composed of patients with pneumoconiosis.
- Dust exposure group: This group is composed of patients exposed to dust.
- Healthy control group: This group is composed of healthy control subjects.

SUMMARY:
The primary objective of this study is to characterize the demographic and clinical features of patients with occupational pneumoconiosis (hereinafter referred to as pneumoconiosis) in China. Secondary objectives include: 1) to describe the natural course of pneumoconiosis; 2) to evaluate the prognosis of pneumoconiosis patients; and 3) to assess complications and comorbidities in pneumoconiosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as pneumoconiosis

Exclusion Criteria:

* Incomplete occupational history information
* Has participated in any interventional clinical research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were selected during physical examinations or during hospitalization from medical organization.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | 3 years
  Pulmonary function tests (PFTs) are utilized to assess the severity of the patient's condition, monitor disease progression, guide therapeutic decision-making, and evaluate prognosis.

SECONDARY OUTCOMES:
Number of patients | 6 years
  The researchers used inclusion/exclusion criteria for screening, and collected the demographic information, clinical symptoms and signs, laboratory tests, treatment, survival and other conditions of the patients who agreed to participate in the program and signed the informed consent, and collected biological specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China